CLINICAL TRIAL: NCT00031642
Title: Phase I/II Study of IDEC-Y2B8 (Zevalin) for Post Transplant Relapses of B-Cell Non-Hodgkin's Lymphoma
Brief Title: Monoclonal Antibody Therapy in Relapsed Non-Hodgkin's After Chemotherapy and Autologous Stem Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0535-00-FB; CDR0000069211 (Registry Identifier: PDQ (Physician Data Query)); NCI-V02-1691 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: rituximab
Radiation: yttrium Y 90 ibritumomab tiuxetan

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and deliver cancer-killing substances to them without harming normal cells. Radiolabeled monoclonal antibodies can locate and deliver radioactive cancer-killing substances.

PURPOSE: Phase I/II trial to study the effectiveness of combining radiolabeled monoclonal antibodies with rituximab in treating patients who have non-Hodgkin's lymphoma that has not responded to high-dose chemotherapy and autologous stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of yttrium Y 90-labeled ibritumomab tiuxetan when administered with rituximab in patients with B-cell non-Hodgkin's lymphoma who have relapsed after high-dose chemotherapy and autologous hematopoietic stem cell transplantation.
* Determine the safety and efficacy of this regimen in these patients.

OUTLINE: This is a dose-escalation study of yttrium Y 90-labeled ibritumomab tiuxetan (IDEC-Y2B8).

* Phase I: Patients receive rituximab IV over 4-6 hours followed by indium In 111-labeled ibritumomab tiuxetan (IDEC-In2B8) IV over 10 minutes on day 0. Patients receive rituximab IV again on day 7 followed by IDEC-Y2B8 IV over 10 minutes.

Cohorts of 3-6 patients receive escalating doses of IDEC-Y2B8 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 3 of 6 patients experience dose-limiting toxicity.

* Phase II: Once the MTD is determined, 58 additional patients are treated at that dose level as in phase I.

Patients are followed at 6 weeks, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 78 patients (20 for phase I and 58 for phase II) will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed B-cell non-Hodgkin's lymphoma (NHL) after high-dose chemotherapy and autologous stem cell transplantation
* Less than 25% bone marrow involvement with NHL as evidenced by unilateral or bilateral biopsy within the past 6 weeks

  o Bone marrow biopsy should demonstrate 15-20% of cellular space occupied by normal hematopoiesis
* CD20 antigen expression in tumor tissue within the past year as evidenced by 1 of the following:

  * Immunoperoxidase stains of tissue showing positive reactivity with L26 antibody
  * Flow cytometry studies
* Measurable disease

  o More than 2 cm bidimensionally
* 19 years of age and over
* Performance status WHO 0-2
* Life expectancy at least 3 months
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 150,000/mm^3
* Bilirubin less than 2.0 mg/dL
* SGOT or SGPT no greater than 2.5 times upper limit of normal (unless due to lymphomatous infiltration of the liver)
* Creatinine less than 2.0 mg/dL
* Fertile patients must use effective contraception during and for 6 months after study therapy
* HIV negative
* At least 4 weeks since prior growth factors
* At least 4 weeks since prior biologic therapy
* At least 4 weeks since any prior cytotoxic chemotherapy (6 weeks for nitrosoureas)
* At least 4 weeks since prior radiotherapy
* Recovered from all prior therapy
* At least 4 weeks since prior immunosuppressants

Exclusion Criteria:

* No active CNS lymphoma
* No HIV- or AIDS-related lymphoma
* No transfusion dependency
* No active obstructive hydronephrosis
* Not pregnant or nursing/negative pregnancy test
* No active infection requiring oral or IV antibiotics
* No human antimurine antibody positivity
* No other major medical problems
* No dependency on hematopoietic growth factors (e.g., epoetin alfa, interleukin-11, filgrastim [G-CSF], or sargramostim [GM-CSF])
* No prior radioimmunotherapy
* No other concurrent biologic therapy of any kind
* No prior fludarabine
* No concurrent chemotherapy
* No concurrent steroids except as maintenance for non-cancerous disease
* No prior pelvic radiotherapy
* No prior radiotherapy to more than 25% of estimated bone marrow reserve
* No concurrent external beam radiotherapy
* No other concurrent investigational drugs
* No other concurrent anti-cancer therapy

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2005-11-01 (Actual); Study Completion 2008-03-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose
Safety and efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, Study Chair — University of Nebraska
Locations (1):
- Eppley Cancer Center at University of Nebraska Medical Center, Omaha, Nebraska, United States